CLINICAL TRIAL: NCT01744691
Title: An Open-label, Single Arm, Multicenter Phase 2 Study of the Bruton's Tyrosine Kinase Inhibitor PCI-32765 (Ibrutinib) in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma With 17p Deletion (RESONATE™-17)
Brief Title: A Multicenter Phase 2 Study of Ibrutinib in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) With 17p Deletion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1117-CA; 2012-004476-19 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-07 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-01

CONDITIONS: Chronic Lymphocytic Leukemia With 17p Deletion; Small Lymphocytic Lymphoma With 17p Deletion
Keywords: CLL; SLL
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ibrutinib (Experimental): All subjects will receive ibrutnib 420 mg (3 x 140-mg capsules) orally once daily.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — All subjects will receive ibrutinib 420 mg (3 x 140-mg capsules) orally once daily.

SUMMARY:
An Open-label, Single arm, Multicenter Phase 2 Study of the Bruton's Tyrosine Kinase Inhibitor ibrutinib in Patients with Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma with 17p Deletion

DETAILED DESCRIPTION:
This is a multicenter, international, open-label, single arm, Phase 2 study designed to evaluate the efficacy and safety of ibrutinib in subjects with relapsed/refractory CLL or SLL with del 17p. All subjects will receive ibrutinib until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Key Inclusion Criteria:

* Documentation of del (17p13.1)
* Must have relapsed or refractory CLL/SLL after receiving at least 1 prior line of systemic therapy.
* Measurable nodal disease by computed tomography (CT)

Key Exclusion Criteria:

* History or current evidence of Richter's transformation or prolymphocytic leukemia
* Prior hematologic stem cell transplantation <6 months from study enrollment or any ongoing GVHD
* Prior exposure to ibrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvina Chu, MD, Study Director — Pharmacyclics LLC.
Locations (55):
- United States (18):
  - Phoenix, Arizona
  - Duarte, California
  - Greenbrae, California
  - La Jolla, California
  - Stanford, California
  - Tampa, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Hackensack, New Jersey
  - New Hyde Park, New York
  - New York, New York
  - Goldsboro, North Carolina
  - Columbus, Ohio
  - Toldedo, Ohio
  - Houston, Texas
- Australia (4):
  - Adelaide
  - Coburg
  - East Melbourne
  - Fremantle
- Belgium (7):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Kortrijk
  - Leuven
  - Roeselare
- Edmonton, Alberta, Canada
- Germany (5):
  - Cologne
  - Dresden
  - Heidelberg
  - Munich
  - Ulm
- New Zealand (2):
  - Auckland
  - Christchurch
- Sweden (3):
  - Gothenburg
  - Lund
  - Stockholm
- Turkey (Türkiye) (5):
  - Ankara
  - Gaziantep
  - Istanbul
  - Izmir
  - Kayseri
- United Kingdom (10):
  - Bournemouth
  - Glasgow
  - Leeds
  - Leicester
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Oxford
  - Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Brien S, Jones JA, Coutre SE, Mato AR, Hillmen P, Tam C, Osterborg A, Siddiqi T, Thirman MJ, Furman RR, Ilhan O, Keating MJ, Call TG, Brown JR, Stevens-Brogan M, Li Y, Clow F, James DF, Chu AD, Hallek M, Stilgenbauer S. Ibrutinib for patients with relapsed or refractory chronic lymphocytic leukaemia with 17p deletion (RESONATE-17): a phase 2, open-label, multicentre study. Lancet Oncol. 2016 Oct;17(10):1409-1418. doi: 10.1016/S1470-2045(16)30212-1. Epub 2016 Sep 13. PMID 27637985
- See also: www.pharmacyclics.com — http://www.pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One hundred forty-five subjects were enrolled and 144 subjects received at least 1 dose of PCI-32765 and constitute the all treated population and the safety analysis set.
Groups:
- Ibrutinib: All subjects received ibrutinib 420 mg (3 x 140-mg capsules) orally once daily.
  Ibrutinib: All subjects received ibrutinib 420 mg (3 x 140-mg capsules) orally once daily.
Period: Overall Study
Arm/Group | Ibrutinib
Started | 144 (Participants who received study treatment)
Completed | 101 (Participants who were on study treatment at the time of the primary analysis)
Not Completed | 43
Not completed — Progressive Disease | 18
Not completed — Unacceptable toxicity, AE or death | 18
Not completed — Withdrawal of consent for treatment | 3
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Population: One hundred forty-five subjects were enrolled and 144 subjects received at least 1 dose of PCI-32765 and constitute the all treated population and the safety analysis set.
Groups:
- PCI-32765: All subjects received PCI-32765 420 mg (3 x 140-mg capsules) orally once daily.
  PCI-32765: All subjects received PCI-32765 420 mg (3 x 140-mg capsules) orally once daily.
Arm/Group | PCI-32765
Number analyzed (Participants) | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.9)
Gender [Count of Participants; unit: Participants]
  Female | 48
  Male | 96

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary objective of this study is to evaluate the efficacy of ibrutinib in terms of ORR according to an Independent Review Committee (IRC). ORR based upon IRC assessment is the proportion of responders in the all treated population. Responders were subjects who achieved partial response (PR) or better, ie, complete response (CR), complete response with incomplete marrow recovery (CRi), nodule partial response (nPR) or PR, per IWCLL 2008 criteria with the clarification for treatment-related lymphocytosis.
Time Frame: The median time on study for all treated participants is 33.3 (range 0.5 - 40.1) months
Population: Efficacy analyses were performed on all 144 treated subjects. The primary analysis (PA) used IRC assessment of efficacy endpoints. In the PA, there were no differences between the IRC and investigator responses. IRC assessment was no longer performed after the PA and the final analysis result report investigator-assessed efficacy outcomes.
Measure: Number (95% Confidence Interval); unit: % of participants with response by PI
Arm/Group | Ibrutinib
Number analyzed (Participants) | 144
% of participants with response by PI | 77.8 [70.3 to 83.8]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: Number of participants who had experienced at least one treatment emergent AE
Time Frame: From first dose of PCI-32765 to within 30 days of last dose for each participant or until study closure
Population: Participants who received at least 1 dose of PCI-32765 and constitute the all treated population.
Measure: Number; unit: participants
Groups:
- PCI-32765: All subjects will receive PCI-32765 420 mg (3 x 140-mg capsules) orally once daily.
  PCI-32765: All subjects will receive PCI-32765 420 mg (3 x 140-mg capsules) orally once daily.
Arm/Group | PCI-32765
Number analyzed (Participants) | 144
participants | 144

ADVERSE EVENTS:
Time Frame: From first dose of PCI-32765 to within 30 days of last dose
Arm/Group | PCI-32765
Serious Adverse Events (participants affected / at risk) | 76/144
Other Adverse Events (participants affected / at risk) | 144/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=144)
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 8
Acute myocardial infarction (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Iritis (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 2
Asthenia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Localised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 21
Urinary tract infection (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Aspergillus infection (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Gastroenteritis clostridial (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lower respiratory tract infection viral (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Lymphadenitis bacterial (Infections and infestations) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Sinusitis fungal (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Varicella zoster virus infection (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Critical illness polyneuropathy (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal infarct (Renal and urinary disorders) | 1
Prostatomegaly (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Trichodysplasia spinulosa (Skin and subcutaneous tissue disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCI-32765 (N=144)
Anaemia (Blood and lymphatic system disorders) | 33
Neutropenia (Blood and lymphatic system disorders) | 29
Increased tendency to bruise (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 21
Spontaneous haematoma (Blood and lymphatic system disorders) | 8
Atrial fibrillation (Cardiac disorders) | 16
Vision blurred (Eye disorders) | 16
Visual acuity reduced (Eye disorders) | 12
Dry eye (Eye disorders) | 11
Lacrimation increased (Eye disorders) | 11
Eye irritation (Eye disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 63
Nausea (Gastrointestinal disorders) | 34
Constipation (Gastrointestinal disorders) | 21
Dyspepsia (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 54
Pyrexia (General disorders) | 31
Oedema peripheral (General disorders) | 28
Chills (General disorders) | 9
Peripheral swelling (General disorders) | 9
Upper respiratory tract infection (Infections and infestations) | 30
Urinary tract infection (Infections and infestations) | 30
Pneumonia (Infections and infestations) | 28
Nasopharyngitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 16
Bronchitis (Infections and infestations) | 14
Cellulitis (Infections and infestations) | 9
Contusion (Injury, poisoning and procedural complications) | 10
Fall (Injury, poisoning and procedural complications) | 8
Weight increased (Investigations) | 20
Weight decreased (Investigations) | 16
Decreased appetite (Metabolism and nutrition disorders) | 28
Hyperuricaemia (Metabolism and nutrition disorders) | 18
Hyponatraemia (Metabolism and nutrition disorders) | 11
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 41
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28
Back pain (Musculoskeletal and connective tissue disorders) | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Headache (Nervous system disorders) | 18
Dizziness (Nervous system disorders) | 14
Peripheral sensory neuropathy (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 12
Depression (Psychiatric disorders) | 10
Anxiety (Psychiatric disorders) | 8
Haematuria (Renal and urinary disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 46
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 23
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Rash erythematous (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 11
Skin lesion (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No